CLINICAL TRIAL: NCT07195071
Title: Feasibility Trial of Combination of Obstetrical Carrier Screening and Hereditary Cancer Screening
Acronym: FOCUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Principal Investigator, Shayan M. Dioun, Assistant Professor of Obstetrics and Gynecology, Division of Gynecologic Oncology, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AAAV8327
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Hereditary Cancer Syndrome
Keywords: obstetrical carrier screening; Pregnant women; prenatal screening; carrier screening; genetic testing; hereditary cancer; hereditary cancer genetic testing
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A: Hereditary cancer testing (Experimental): Hereditary Cancer screenings testing and Obstetric Cancer Screening
  Interventions: Device: Natera empower comprehensive hereditary cancer panel; Device: Obstetrical carrier screening
- Arm B: No hereditary caner testing (Active Comparator): Obstetric Cancer screening test only
  Interventions: Device: Obstetrical carrier screening

INTERVENTIONS:
Device: Natera empower comprehensive hereditary cancer panel — Natera Empower Comprehensive Hereditary Cancer Panel to screen for hereditary cancers
  Arms: Arm A: Hereditary cancer testing
Device: Obstetrical carrier screening — Obstetrical carrier screening for genetic conditions

SUMMARY:
The investigators hypothesize that preconception and pregnancy may be a feasible and effective time to offer inherited cancer risk screening. This study will assess interest in cancer genetic testing among patients receiving routine prenatal care or preconception care. The goal is to evaluate the acceptability of hereditary cancer testing when offered alongside standard prenatal genetic screening. The study will also explore whether universal screening in this population could support early cancer prevention

DETAILED DESCRIPTION:
In this prospective trial, a clinician in the department of OBGYN will meet with preconception/pregnant patients who are undergoing obstetrical carrier screening (OCS) at Columbia University affiliated OBGYN clinics to review the options for concurrent hereditary cancer screening (HCS). If interested in the study, the patient will be contacted by a study coordinator and offered participation in the study. The patients will have counseling on potential risks and benefits of genetics testing and have OCS performed per standard of care protocols. This consultation will include collection of comprehensive personal and family history to generate a cancer genetic risk assessment. The patient will be counseled based on their cancer genetic risk assessment, whether or not National Comprehensive Cancer Network (NCCN) guidelines for cancer risk assessment are met and the resulting anticipated cost. The patient will be offered additional consultation with a genetic counselor and/or a Natera financial representative if desired for further counseling. If the patient decides to proceed with HCS, the Natera Empower Hereditary Cancer Panel will be drawn at the time of the OCS panel blood draw and sent to Natera for processing. OCS results will be sent separately and reported to the patient based on standard protocols. Patients that have HCS panels sent will be notified of their results by a genetic counselor from Columbia University's Department of OBGYN and standard of care post test counseling/referrals made.

The study team will evaluate patient acceptance of testing and the patient experience, via validated surveys conducted at time of testing. The study team will evaluate if patient sociodemographic characteristic (e.g. age, parity, race, ethnicity, medical history, family history) are associated with patient acceptance of the combined OCS/HSC panel. Patients that elect to undergo HCS panel will also complete the Regret About Healthcare Decisions Survey after receiving their HCS results. Participation in surveys is encouraged but not mandatory. All patient demographics, survey screens and results will be stored in a secure online database maintained by Columbia University's Department of OBGYN. This data will be entered and maintained by study personal at Columbia University. Patients enrolled in the study will be invited to participate in an interview conducted by telephone at times convenient for them. Interviews will be conducted by language-concordant, trained qualitative experts. Interviews will be recorded and transcribed. Participation in the interview is not mandatory.

Patients that completed HCS and had a mutation that resulted in a recommendation for clinical follow up (e.g. BRCA 1/2 mutation with recommendation for breast screening) will be contacted by telephone at 18 months and asked whether they completed the medical follow-up prompted by HCS results. Participation in this follow-up is not mandatory.

ELIGIBILITY:
Inclusion criteria:

* Age: 18 years - 55 years
* Patients receiving obstetrical-related care at a CUMC-affiliated enrollment site
* Patients who have elected to undergo OCS with the CUMC-affiliated obstetrics provider
* Patients with prior OCS but planned to repeat OCS are eligible
* Patients can speak and read in English or Spanish

Exclusion criteria:

* Patients who have previously completed a multigene hereditary cancer syndrome panel
* Patients that have a hematologic cancer or hematologic pre-cancer
* Patients who have a history of an autologous bone marrow transplant

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Complete Both HCS and OCS | Approximately at the end of recruitment, expected at 2 years
  The percent of patients who complete hereditary cancer screening (HCS) when offered in addition to routine obstetrical carrier screening (OCS) during preconception and obstetrical-related care.

SECONDARY OUTCOMES:
Score on Regret About Healthcare Decisions survey | 2 to 6 months after enrollment
  Participant experience with combined HCS and OCS will be assessed using a validated Regret About Healthcare Decisions Survey. The minimum score is 0 (lowest regret) to 100 (highest regret).
Score on Regret About Healthcare Decisions Survey among pregnant participants | Approximately at the end of recruitment, expected at 2 years
  Assessment of participant experience with combined OCS and HCS in pregnant participants using Regret About Healthcare Decisions Survey and qualitative interviews. The minimum score is 0 (lowest regret) to 100 (highest regret).
Score on Regret About Healthcare Decisions Survey among nonpregnant participants | Approximately at the end of recruitment, expected at 2 years
  Assessment of participant experience with combined OCS and HCS in nonpregnant participants using Regret About Healthcare Decisions Survey and qualitative interviews. The minimum score is 0 (lowest regret) to 100 (highest regret).
Hereditary cancer screening results | Approximately at the end of recruitment, expected at 2 years
  Number of pathologic variants identified by hereditary cancer screening.
Percentage of High-Risk Participants Utilizing Guideline-Based Cancer Mitigation Strategies | 18 months after enrollment
  Among participants who complete both HCS and OCS and are identified as being at elevated cancer risk, this measure captures the percentage who undergo one or more guideline-based cancer mitigation strategies, such as mammogram, breast MRI, or colonoscopy.
Percentage of Participants Who Complete Both HCS and OCS during pregnancy | Approximately at the end of recruitment, expected at 2 years
  The percent of patients who complete hereditary cancer screening (HCS) when offered in addition to routine obstetrical carrier screening (OCS) while pregnant.

CONTACTS AND LOCATIONS:
Overall Officials: Shayan Dioun, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided